CLINICAL TRIAL: NCT06754683
Title: The Effect of Self-Compassion-Based Psycho-Education on Nursing Students' Self-Compassion, Stress, Resilience, and Psychological Well-Being
Brief Title: The Effect of Self-Compassion Interventions on Nursing Students' Stress, Resilience, and Psychological Well-Being
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Samineh Esmaeilzadeh, Principal Investigator, Near East University, Turkey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NEU/2024/128-1889
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: To Determine the Impact of Self-compassion Intervention
Keywords: Self-compassion; Stress; Resilience; Psychological Well-being; Nursing Students
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: After the study period for the intervention group, the control group will be switched to the intervention group for the same period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassion based psycho-education intervention (Experimental): 8-week Self-compassion based psycho-education intervention
  Interventions: Behavioral: 8 weeks Self-compassion based psycho-education
- Wait-list control group (No Intervention): A pre-test will be conducted in the first week and the post-test in the 8th week.

INTERVENTIONS:
Behavioral: 8 weeks Self-compassion based psycho-education — The Self-compassion psychoeducational intervention will be utilized as the intervention in this study will be delivered by the first investigator and supervised by the Principal investigator, who has experience in mindfulness and self-compassion practices. It will consist of eight weekly 1.5 hours of face-to-face sessions and 1 hour each week of online sessions. Each session will be according to a specific topic that will cover the objectives of the study, incorporating the concept of self-compassion interventions based on the research literature and input from experts in the field, taking into consideration the needs of the participants. Participants will be required to have at least 80% of attendance for intervention completion.
  Arms: Self-compassion based psycho-education intervention

SUMMARY:
The study aims to determine the impact of self-compassion-based psycho-education on supporting nursing students in managing stress, improving their resilience, and enhancing their self-compassion and psychological well-being (PWB). Self-compassion involves being kind to oneself during challenging times; it provides practical tools and knowledge to enhance personal growth and resilience. By participating in this program, nursing students may learn strategies to improve their coping with the pressure of studies, build emotional strength, and improve their psychological well-being. The study will measure the participants' levels of self-compassion, stress, resilience, and psychological well-being using a validated questionnaire before and after participation in the program and compare them to determine the program's impact on the abovementioned variables.

DETAILED DESCRIPTION:
The below standard operating procedures will be used to make sure that the study's patient recruitment, data collection, data management, data analysis, and reporting of adverse events are all done consistently and accurately in line with ethical standards: The inclusion and exclusion criteria, which specify the eligibility criteria, will guide the recruitment of participants. The recruitment process will use various student communication channels, such as emails, social media, and classroom announcements, to invite participants to the study. The investigators will provide study details to the participants before obtaining informed consent; demographic information about the participants and their recruitment status will be kept in secure folders. The investigators will use validated instruments before and after the intervention to measure self-compassion, stress, resilience, and psychological well-being, as approved by the ethics committee and data quality control procedures. The self-compassion-based psychoeducation will be delivered according to the protocol approved by the ethics committee. Participants' identities will be confidential and kept in secure password-protected systems for storing data; the investigators will conduct regular audits during data entry to ensure consistency and accuracy. Statistical Package software for social sciences, version 25, will be used for analysis as planned in collaboration with a statistical analysis expert to ensure accurate interpretation of the results. The participants will be given information and contact information of the investigators to report adverse events, such as any unexpected psychological distress during or after the program. The research team will document, follow up with the participants, and refer them to the university counseling center if necessary.

Using G power, the researchers carried out a-priori power analysis to determine the sample for the study since the literature search that the investigators conducted did not show any interventional study that assessed the effect of the self-compassion psycho-education intervention on self-compassion, stress, resilience, and psychological well-being, the investigators draw reference to methods used by Yip and Tong (2019) when conducting study, the researchers used the effect size results of self-compassion intervention meta-analysis of Zessin et al. (2015); the analysis found large effect size (g = 0.90) between self-compassion and well-being. The sample size required for 90% (1-β = 0.90) power at α=0.05 level for the assumption that the effect size will be large (d=0.90) in the study was calculated as 54 participants, 27 for each group, using G*Power 3.1.9.2 software, t-tests - repeated measures difference between two independent means analysis: A priori: Compute required sample size Input: Effect size d = 0.9, α err prob = 0.05, Power (1-β err prob) = 0.90, allocation ratio N2/N1 Output: noncentrality parameter λ = 3.30, Critical t = 2.00, df = 52, Total sample size = 54, actual power = 0.90. Considering the withdrawal rate (attrition rate) of 17% in a study of self-compassion intervention by Yang et al. (2024), the researchers calculated 17% of the calculated sample in this study (54/100 = 0.54 * 17 = 9.18, approximately 10). Therefore, the calculated sample size (54) and the addition of the computed attrition rate (10) will give a total of 64 participants (32 each for the intervention and the control group). Subjects will be recruited through convenience sampling.

To ensure the integrity and validity of results, the investigators will use validated data collection tools, conduct periodic checks during data collection, and maintain regular communication and simple explanations to participants to encourage complete and accurate responses. Investigators will regularly check the collected data for completeness and the data entries for further review and possibly record the type and extent of missing data in a log for transparency. Depending on the type of data missing, the investigators will handle it appropriately through coding, imputation technique, or exclusion criteria; the investigators will assess the pattern of the missing data and undertake sensitivity analysis to examine the impact of missing data on results and validate conclusions; the investigators will report all the above if it occurs to ensure transparency in handling missing data without altering participants' responses.

Evaluation of Data: All data will be analyzed using the study's Statistical Package for the Social Sciences (SPSS) version 25. Descriptive statistics (frequencies, percentages, mean, and standard deviation) will be used to describe the demographic data and summary of the scores of the state self-compassion scale long form (SSCS-L), stress, resilience, and PWB. For the impact of the intervention, a normality test will be conducted using the Kolmogorov-Smirnov test, and an appropriate statistical test will be applied after the test; for instance, an independent t-test will be utilized for between-group comparisons if the test satisfies the assumptions of a parametric independent t-test. The alternative nonparametric test (Mann-Whitney U Test) will be used if the assumption is unmet. For within-group comparisons, if the data satisfy the assumption of the parametric test, paired t-tests will be applied to assess changes in the intervention group between the pre-test and post-test, as well as those of the control group. The significance level will be set at p < 0.05; if the assumption of the parametric test (paired t-tests) is not met, a nonparametric alternative (Wilcoxon signed rank test) will be used, and the significance level will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* International students of Nursing Faculty
* The participants should be able to communicate effectively using the English language.
* Participants did not participate in self-compassion -based training before
* The subject has commenced clinical posting and experience.
* Participants with low self-compassion score in the preliminary survey

Exclusion Criteria:

* Participants receiving psychotherapy
* Participants who are currently enrolled in any online or face-to-face stress management training or course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in self-compassion score as measured by state self-compassion scale (SSCS-L) | Baseline, 8 Weeks
  Self-compassion score as measured by the SSCS-L, is a 5 rating scale with 1= not at all true for me to 5= Very true for me with a total of 18 items that can assess total (composite) self-compassion score as well as the six (kindness, self-judgment, mindfulness, over-identification, common humanity and isolation) individual elements of self-compassion. To compute a total state self-compassion score: the investigators will take the mean of each subscale, to compute a total mean (the average of the six subscale means as suggested by the scale authors). The score cut-off point is 1.0-2.49 to be low, 2.5-3.5 to moderate, and 3.51-5.0 to be high. When examining subscale scores, higher scores on the self-judgment, isolation, and over-identification scale indicate less self-compassion before reverse-coding, and more self-compassion after reverse coding.
Psychological well-being score as measured by brief inventory of thriving scale (BITS) | Baseline, 8 Weeks
  Psychological well-being score as measured by brief inventory of thriving scale, it is a 5 Likert rating scale with 1= totally disagree to 5= totally agree with a total of 10 items. The scores cut off point is 1.0-2.49 to be low, between 2.5-3.5 to be moderate, and 3.51-5.0 to be high.

SECONDARY OUTCOMES:
Change in stress score as measured by student nurse stress index scale (SNSI) | Baseline, 8 Weeks
  Stress as measured by student nurse stress index scale, it is a 5 Likert rating scale with 1= Not stressful to 5= Extremely stressful with a total of 22 items. The SNSI is scored on a continuum, from not stressful (22) to extremely stressful (110)
Change in resilience score as measured by Connor-Davidson-Resilience-Scale (CD-RISC-10 scale). | Baseline, 8 Weeks
  Resilience as measured by CD-RISC-10 scale, it is a 5 rating scale with 0= not true at all to 4= true nearly all the time, with a total of 10 items. The total of the rating will give a composite score that ranges from 0 to 40. Higher score rating will represent greater resilience while lower score will indicate low resilience.

CONTACTS AND LOCATIONS:
Overall Officials: SAMINEH ESMAEILZADEH, PhD, Principal Investigator — Near East University, Turkey
Locations (1):
- Near East University, Turkey, Yakın Doğu Bulvarı, Mersin 10, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) sharing plan in this study includes a detailed study protocol, available upon request after the publication of the results. A statistical plan outlining the methods and analysis used to address objectives will be available after the publication of the results in peer-reviewed journal. The unidentified consent form explaining the study purpose, procedures, possible risks, and participants' rights will be available upon request and institutional review board (IRB) approval. After completing the studies, the analytic code for data cleaning and statistical analysis will be made available upon reasonable request. IPD will be shared within 6-12 months after the publication of results in a peer-reviewed journal; it will also be shared through secure online repositories (clinicalTrials.gov) and Near East University (NEU) library repository; data access requires a data use agreement and a summary of research objectives, evaluated for ethical compliance.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be shared within 6-12 months after the publication of results in a peer-reviewed journal
Access Criteria: Researchers and participants will be able to access data on all collected IPD and all IPD that underlie results in the result publication of this study

REFERENCES:
- [Background] Klainin-Yobas P, Vongsirimas N, Ramirez DQ, Sarmiento J, Fernandez Z. Evaluating the relationships among stress, resilience and psychological well-being among young adults: a structural equation modelling approach. BMC Nurs. 2021 Jul 5;20(1):119. doi: 10.1186/s12912-021-00645-9. PMID 34225712
- [Background] Kilic A, Hudson J, McCracken LM, Ruparelia R, Fawson S, Hughes LD. A Systematic Review of the Effectiveness of Self-Compassion-Related Interventions for Individuals With Chronic Physical Health Conditions. Behav Ther. 2021 May;52(3):607-625. doi: 10.1016/j.beth.2020.08.001. Epub 2020 Aug 13. PMID 33990237
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Huang, J., Lin, K., Fan, L., Qiao, S., & Wang, Y. (2021). The effects of a self-compassion intervention on future-oriented coping and psychological well-being: A randomized controlled trial in Chinese college students. Mindfulness, 12, 1451-1458. https://doi.org/10.1007/s12671-021-01614-8
- [Background] Jones, M. C., & Johnston, D. W. (1999). The derivation of a brief Student Nurse Stress Index. Work & Stress, 13(2), 162-181. https://doi.org/10.1080/026783799296129
- [Background] Neff, K. D., Tóth-Király, I., Knox, M. C., Kuchar, A., & Davidson, O. (2021). The Development and Validation of the State Self-Compassion Scale (Long-and Short Form). Mindfulness, 12(1), 121-140. https://doi.org/10.1007/s12671-020-01505-4
- [Background] Su R, Tay L, Diener E. The development and validation of the Comprehensive Inventory of Thriving (CIT) and the Brief Inventory of Thriving (BIT). Appl Psychol Health Well Being. 2014 Nov;6(3):251-79. doi: 10.1111/aphw.12027. Epub 2014 Jun 12. PMID 24919454
- [Background] Tung, L. N. (2020). Using Mindful Self-Compassion (MSC) as a Strategy to Reduce Stress and Develop Self-Compassion in Nursing Students (Order No. 27837495). Available from ProQuest Dissertations & Theses Global. (2458948204). https://www.proquest.com/dissertations-theses/using-mindful-self-compassion-msc-as-strategy/docview/2458948204/se-2
- [Background] Yang Z, Tse MMY, Huang H, Fang H, Chung JWY, Chong DYK, Wong TKS. Evaluating the feasibility and preliminary effects of an online compassion training program for nursing students: A pilot randomized controlled trial. Int J Nurs Sci. 2024 Aug 12;11(4):421-428. doi: 10.1016/j.ijnss.2024.08.007. eCollection 2024 Sep. PMID 39830914